CLINICAL TRIAL: NCT04102852
Title: The Role of Lactobacillus Rhamnosus GG (ATCC 53103) in the Modulation of the Inflammatory Process in the Mucosa of Ulcerative Colitis (UC) Patients With Mild-moderate Clinical Activity
Brief Title: Lactobacillus Rhamnosus GG (ATCC 53103) in Mild-moderately Active UC Patients
Acronym: LGGinUC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: San Giovanni Addolorata Hospital (Other)
Collaborators: Onlus S. Andrea (Unknown)
Responsible Party: Principal Investigator, Cristiano Pagnini, Principal Investigator, San Giovanni Addolorata Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LGG/UC/001
Record Dates: First submitted 2019-09-17; First posted 2019-09-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis Chronic Mild; Ulcerative Colitis Chronic Moderate
Keywords: probiotic; Lactobacillus rhamnosus GG; ATCC 53103; cytokines; adhesion
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients do not know if the LGG dose they a taking is the "regular" ot the "double" dose The investigator that assess the parameters at the end of the treatment is different from the investigator that examined the patient at the pre-treatment visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LGG regular dose (Experimental): Patients taking LGG 1.2 × 10^10 CFU/day, 2 capsules a day, for 1 month
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG ATCC 53103
- LGG double dose (Experimental): Patients taking LGG 2.4 × 10^10 CFU/day, 4 capsules a day, for 1 month
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG ATCC 53103

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG ATCC 53103 — probiotic administration at two different doses for 1 month

SUMMARY:
This study is a randomized double-blind clinical trial that intends to evaluate the efficacy and safety of LGG administration at two different doses, for 1 month, in ulcerative colitis (UC) patients with mild-moderate disease activity in therapy with oral mesalamine. Efficacy of therapy will be evaluated by clinical (Clinical Mayo score, quality of life assessment), endoscopic (Endoscopic Mayo score), histological, biochemical (white cell count, C-reactive protein), and molecular (mucosal colonization of the bacteria, pro- and anti-inflammatory cytokines measurement) parameters. UC patients with mild-moderately active disease despite oral treatment with mesalamine will be assessed at baseline for clinical, endoscopic, histologic inflammatory activity. After a wash-out period of 4 weeks of mesalamine, patients will be randomized to assume a regular (LGG 1.2 × 10^10 Colony Forming Units (CFU)/day, 2 capsules a day) or a double (LGG 2.4 × 10^10 CFU/day, 4 capsules a day) dose of LGG for 1 month. At the end of the treatment, clinical, endoscopic, and histologic inflammatory activity will be evaluated and compared to pre-treatment data. Adhesion and molecular effect of LGG will be also evaluated. Safety will be assessed by weekly phone calls and with direct physical examination at the end of the study period.

DETAILED DESCRIPTION:
Probiotic bacteria have been proposed as therapeutic option in several pathologic conditions, but their utilization is often not evidence-based driven. In inflammatory bowel disease (IBD), consistent heterogenity exists among published clinical studies. Aim of the present clinical study is to evaluate the effect of Lactobacillus rhamnosus GG (LGG), the probiotic bacteria most extensively investigated, with solid safety data and proven anti-inflammatory effect in experimental models, in ulcerative colitis (UC) patients, with a rigorous methodology, a well defined protocol, and with relevant outcomes clearly set.

This study is a randomized double-blind clinical trial that intends to evaluate the efficacy and safety of LGG administration at two different doses, for 1 month, in UC patients with mild-moderate disease activity in therapy with oral mesalamine.The eligible patients will be identified by a screening visit (T-1), with consideration of inclusion and exclusion criteria, and informed consent will be signed. Then the patients will have a 4 weeks wash-out period, when oral mesalamine will be suspended, and biochemical tests [total blood count, C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), and serum protein electrophoresis], and endoscopic examination with biopsies will be performed. The patients will be then evaluated again prior to the randomization to regular or double dose group (T0), and clinical activity and quality of life will be assessed. Patients will be randomized to assume a regular (LGG 1.2 × 10^10 CFU/day, 2 capsules a day) or a double (LGG 2.4 × 10^10 CFU/day, 4 capsules a day) dose of LGG for 1 month. After 4 weeks of treatment, patients will be re-evaluated (T1), with physical examination and interview, and rectum-sigmoidoscopy with biopsies will be performed. The patients will then be allowed to assume the therapy they were taking at T-1 visit (mesalamine), and will be assessed for the last time after 4 weeks after treatment completition (T2), with physical examination and interview. Efficacy of therapy will be evaluated by comparison of clinical, endoscopic, histological, biochemical and molecular data, pre- and post-treatment (T1 vs. T0). Randomization of patients in the groups will be performed by a computer-generated randomization list, in a double blind fashion. Clinical activity will be evaluated by Clinical Mayo Score calculation. Quality of life will be evaluated by specific validated tests. Endoscopic activity will be evaluated by Endoscopic Mayo Score calculation, by an endoscopist blinded to clinical data of patients. Histologic activity will be evaluated by expert anatomopathologists, by means of Geboes score. Molecular activity of LGG will be evaluated by assessment of bacteria adhesion to the colonic mucosa, measured by real-time(RT)-Polymerase Chain Reaction (PCR) with specific primers on total DNA extracted by bioptic samples (as already described), and by quantification of expression of pro- and anti-inflammatory cytokines, before and after probiotic treatment, by means of RT-PCR on total RNA extracted from bioptic samples (as already described).

Safety of LGG treatment will be assessed by weekly phone calls to the patients, in order to investigate the unexpected occurence of side-effects, and with direct physical examination and biochemical tests at the end of the study period (T1). Possible LGG translocation will be evaluated by RT-PCR with specific primers on total DNA extracted from peripheral blood collected from patients at the end of treatment (T1).

ELIGIBILITY:
Inclusion Criteria:

* firm diagnosis of UC (clinical, endoscopic and histological criteria) from at least 1 year
* mild-moderate clinical activity (Clinical Mayo score 2-4)
* patient taking oral mesalamine
* Informed consent obtained and signed at the screening visit (T-1)

Exclusion Criteria:

* Pregnant women
* Serious co-morbidities (i.e. autoimmune pathologies, cancer, chronic infectious conditions, immunocompromised patients)
* Patients at first diagnosis of UC
* Patients with current immunosuppressive and/or biologic therapy for IBD, or who had immunosuppressive and/or biologic therapy for IBD in the last year
* Patients with current oral and/or topical steroid therapy, or who had oral steroid therapy for disease flare in the last 6 months
* Patients with current topical UC therapy (suppositories, enemas, foams)
* Patients with current antibiotic/probiotic therapy, or who had antibiotic/probiotic therapy in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Clinical Mayo Score after treatment [Efficacy] | 1 month
  Improvement of clinical inflammatory activity (Clinical Response) evaluated by reduction of Clinical Mayo Score at the end of the treatment comparing to pre-treatment value
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | every week, through 1 month
  Recording and description of any side effect possibly related to probiotic administration

SECONDARY OUTCOMES:
Mucosal Adhesion of LGG to Colonic Mucosa | 1 month
  Effective LGG colonization in colonic mucosa as measured by real-time PCR detection of LGG in bioptic samples of colon of LGG treated patients at the end of the treatment
Quality of Life Improvement | 1 month
  Improvement of QoL parameters as measured and assessed by Short Form-36 Health Survey (SF-36), before and after probiotic treatment. The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state. The final score is generated by a formula that combines the different domains' score, and expressed by a score with a 0 to 100 range,with a higher score defining a more favorable health state

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Pagnini, MD, PhD, Principal Investigator — S.Giovanni Addolorata Hospital; Gianfranco Delle Fave, MD, Study Director — Onlus S. Andrea
Locations (1):
- S. Giovanni Addolorata Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pagnini C, Corleto VD, Martorelli M, Lanini C, D'Ambra G, Di Giulio E, Delle Fave G. Mucosal adhesion and anti-inflammatory effects of Lactobacillus rhamnosus GG in the human colonic mucosa: A proof-of-concept study. World J Gastroenterol. 2018 Nov 7;24(41):4652-4662. doi: 10.3748/wjg.v24.i41.4652. PMID 30416313
- [Result] Pagnini C, Martorelli M, Lanini C, Delle Fave G. Development of an Ex Vivo Organ Culture Technique to Evaluate Probiotic Utilization in IBD. J Clin Gastroenterol. 2016 Nov/Dec;50 Suppl 2, Proceedings from the 8th Probiotics, Prebiotics & New Foods for Microbiota and Human Health meeting held in Rome, Italy on September 13-15, 2015:S179-S182. doi: 10.1097/MCG.0000000000000698. PMID 27741170
- [Result] Derwa Y, Gracie DJ, Hamlin PJ, Ford AC. Systematic review with meta-analysis: the efficacy of probiotics in inflammatory bowel disease. Aliment Pharmacol Ther. 2017 Aug;46(4):389-400. doi: 10.1111/apt.14203. Epub 2017 Jun 27. PMID 28653751
- [Derived] Pagnini C, Di Paolo MC, Urgesi R, Pallotta L, Fanello G, Graziani MG, Delle Fave G. Safety and Potential Role of Lactobacillus rhamnosus GG Administration as Monotherapy in Ulcerative Colitis Patients with Mild-Moderate Clinical Activity. Microorganisms. 2023 May 24;11(6):1381. doi: 10.3390/microorganisms11061381. PMID 37374884